CLINICAL TRIAL: NCT03172312
Title: Clinical Utility of Intraoperative Parathyroid Scores System in Thyroidectomy
Acronym: IPSS
Status: Completed | Type: Observational
Sponsor: Fujian Medical University (Other)
Responsible Party: Principal Investigator, wangbo, chairmen of thyroid surgery, Fujian Medical University
Other Study IDs: IPSSforZHAO
Record Dates: First submitted 2017-05-29; First posted 2017-06-01 (Actual); Last update posted 2017-06-01 (Actual); Status verified 2017-05

CONDITIONS: Intraoperative Parathyroid Scores System
Keywords: Intraoperative Parathyroid Scores System; total thyroidectomy; thyroid cancer; hypoparathyroidism; prediction
MeSH Terms: conditions — Thyroid Neoplasms; Hypoparathyroidism

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Total thyroidectomy: Patients need to do total thyroidectomy According to guidelines
  Interventions: Procedure: Different range of thyroid surgery
- Hemithyroidectomy: Patients need to do Hemithyroidectomy According to guidelines
  Interventions: Procedure: Different range of thyroid surgery

INTERVENTIONS:
Procedure: Different range of thyroid surgery — Observe and record parathyroid status during thyroid surgery

SUMMARY:
Ready to establish the Intraoperative Parathyroid Scores System (IPSS) for thyroidectomy and study the clinical value of Intraoperative Parathyroid Scores System for thyroidectomy.

DETAILED DESCRIPTION:
IPSS includes transplantation Parathyroid Scores and in situ Parathyroid Scores, the investigators will establish the Intraoperative Parathyroid Scores System by parathyroid size and Blood supply, and recording IPSS, according to certain rules. Parathyroid hormone and calcium were test in d0, d1, d14, d60 post operation. The correlation between Intraoperative Parathyroid Scores and PTH calcium were calculated, and ROC curve and logistic regression were tested for the prediction value.

ELIGIBILITY:
Inclusion Criteria:

1. postoperative pathology confirmed as thyroid papillary carcinoma;
2. for the first time to undergo thyroid surgery, no history of neck surgery and external radiotherapy;
3. preoperative serum calcium, parathyroid hormone levels were normal;
4. intraoperative and postoperative clinical data integrity, standardized follow-up patients;
5. parathyroid is a tumor violation.

Exclusion Criteria:

1. serious underlying disease;
2. age greater than 60 years of age or combined with arteriosclerotic disease;
3. patients with postoperative loss;
4. patients with parathyroid disease.

Max Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients who need thyroid surgery
Sampling Method: Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2014-01-01 (Actual); Primary Completion 2016-12-31 (Actual); Study Completion 2016-12-31 (Actual)

PRIMARY OUTCOMES:
transplantation Parathyroid Scores correlated with transplanted parathyroid function | 2014-2016
  relation with transplantation Parathyroid Scores and transplanted parathyroid hormone
the value of IPSS and in situ Parathyroid Scores | 2014-2016
  relation with Intraoperative Parathyroid Scores and in situ Parathyroid Scores
predicted function of IPSS | 2014-2016
  IPSS and in suit PSS be recoded and D1，D14 PTH Ca2+ were tested
value of IPSS in low PTH patients | 2014-2016
  IPSS and in suit PSS be recoded and D1，D14 PTH Ca2+ were tested

SECONDARY OUTCOMES:
value of IPSS for Surgeon and patient | 2014-2016
  description the clinic value

CONTACTS AND LOCATIONS:
Locations (1):
- Wen-xin ZHAO, Fuzhou, Fujian, China

IPD SHARING:
Plan to Share IPD: No